CLINICAL TRIAL: NCT03791944
Title: 3DV+TPS Applied to Radiotherapy for Nasopharyngeal Carcinoma - a Randomized, Single-blind, Multi-center Clinical Study
Brief Title: 3DV+TPS Applied to Radiotherapy for Nasopharyngeal Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Deputy director, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XQonc-010
Record Dates: First submitted 2018-12-31; First posted 2019-01-03 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Nasopharynx Cancer; Radiotherapy
Keywords: nasopharynx cancer; Radiotherapy
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 3DV+TPS/VARIAN (Experimental): Use 3DV+TPS to map targets and develop treatment plans. The intervention is 3DV+TPS and VARIAN.
  Interventions: Device: 3DV+TPS/VARIAN
- TPS/VARIAN (Active Comparator): Use imported Varian TPS to map targets and develop treatment plans.
  Interventions: Device: TPS / VARIAN
- 3DV+TPS/ Domestic accelerator (Experimental): Use 3DV+TPS to map targets and develop treatment plans.
  Interventions: Device: 3DV + TPS / Domestic Accelerator
- TPS/ Domestic accelerator (Active Comparator): Adopt domestic TPS hook target and develop treatment plan.
  Interventions: Device: TPS / Domestic Accelerator

INTERVENTIONS:
Device: 3DV+TPS/VARIAN — Use imported 3DV+TPS to map targets and develop treatment plans
  Arms: 3DV+TPS/VARIAN
Device: TPS / VARIAN — Use imported TPS to map targets and develop treatment plans
  Arms: TPS/VARIAN
Device: 3DV + TPS / Domestic Accelerator — Use domestic 3DV+TPS to delineate target areas and develop treatment plans
  Arms: 3DV+TPS/ Domestic accelerator
Device: TPS / Domestic Accelerator — Use domestic TPS to map targets and develop treatment plans
  Arms: TPS/ Domestic accelerator

SUMMARY:
Verify that 3DV+TPS is non-inferior compared to existing imported TPS and superior to existing domestic TPS.

DETAILED DESCRIPTION:
The main purpose of the study was to verify that 3DV+TPS is non-inferior compared to existing imported TPS and superior to existing domestic TPS. A total of 100 patients were enrolled. The primary endpoint of the study was the objective response rate (ORR), and the secondary endpoint was the local control rate and the incidence of treatment-related side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Consolidate other serious diseases that affect quality of life or treatment;
2. Reluctant to actively cooperate with the investigator;
3. Mergers with distant transfers;
4. Patients who have undergone head and neck surgery and radiotherapy;
5. Subjects who are affected by the disease who sign a written informed consent or follow the study procedure; or who are unwilling or unable to comply with the research requirements.
6. Those who have a history of psychotropic substance abuse who are unable to quit or have a mental disorder;
7. Participated in other clinical trials of anti-tumor drugs within 4 weeks before enrollment;
8. Pregnant or lactating women;
9. The investigator judges other conditions that may affect the clinical study and the outcome of the study.

Exclusion Criteria:

1. Those who did not follow the protocol.
2. The subject is aggravated or has a serious adverse reaction.
3. The subject himself requested to withdraw from the trial.
4. The patient is lost to follow-up or died.
5. The researcher believes that there is reason to withdraw

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 3 months follow-up after treatment
  Objective Remission Rate (ORR) is equal to complete remission (CR) + partial remission (PR)

SECONDARY OUTCOMES:
Local control rate | 3 months follow-up after treatment
  Local control means that the tumor does not increase in imaging, but if the tumor does not increase, the patient with increased symptoms after treatment is not included in the local control range.
incidence of treatment-related side effects | 3 months follow-up after treatment
  Incidence of related side effects during disease treatment

CONTACTS AND LOCATIONS:
Locations (1):
- the second affiliated hospital of Army medical university, Chongqing, Chongqing Municipality, China